CLINICAL TRIAL: NCT01115673
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Safety and Efficacy Study of Acetaminophen 1000 mg and Acetaminophen 650 mg in Post Operative Dental Pain
Brief Title: To Evaluate the Safety and Efficacy of Acetaminophen 650 mg and 1000mg in Dental Pain After Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McNeil Consumer Healthcare Division of McNEIL-PPC, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACEPAI2001
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ACE-1000 (Experimental): 1000 mg Acetaminophen Caplet
  Interventions: Drug: Acetaminophen
- ACE-650 (Active Comparator): 650 mg Acetaminophen Caplet
  Interventions: Drug: Acetaminophen
- ACE-0 (Placebo Comparator): 0 mg Acetaminophen Caplet
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen Caplet - single dose
  Other Names: Tylenol
  Arms: ACE-1000; ACE-650
Drug: Placebo Control — 0 mg Caplet - single dose
  Other Names: Control
  Arms: ACE-0

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of acetaminophen 650 mg and acetaminophen 1000 mg in dental surgery.

DETAILED DESCRIPTION:
This trial is to assess the relative efficacy of acetaminophen 1000 mg versus acetaminophen 650 mg over a six-hour period, in subjects experiencing at least moderate post-operative dental pain.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 16 and less than 51 years of age
* Must weigh at least 100 lbs with a body mass index of at least 18 and less than 30
* Must have up to four of their back teeth (third-molars) pulled

Exclusion Criteria:

* Cannot be allergic to acetaminophen (Tylenol)
* Cannot be pregnant (or planning to be pregnant) or nursing a baby
* Cannot have any other medical conditions that the investigator determines might compromise your safety or the study results

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 540 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Qi, M.D., Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Qi DS, May LG, Zimmerman B, Peng P, Atillasoy E, Brown JD, Cooper SA. A randomized, double-blind, placebo-controlled study of acetaminophen 1000 mg versus acetaminophen 650 mg for the treatment of postsurgical dental pain. Clin Ther. 2012 Dec;34(12):2247-2258.e3. doi: 10.1016/j.clinthera.2012.11.003. Epub 2012 Nov 28. PMID 23200183

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Started | 239 | 241 | 60
Completed | 239 | 241 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACE-1000 | ACE-650 | ACE-0 | Total
Number analyzed (Participants) | 239 | 241 | 60 | 540
Age Continuous [Mean (Standard Deviation); unit: years] | 18.5 (2.24) | 18.3 (1.96) | 18.1 (2.02) | 18.4 (2.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 120 | 31 | 282
  Male | 108 | 121 | 29 | 258
Region of Enrollment [Number; unit: participants]
  United States | 239 | 241 | 60 | 540

OUTCOME MEASURES:

1. Primary Outcome: Overall Analgesic Efficacy - Sum of Pain Intensity Difference and Pain Relief Scores Over Six Hours (SPRID6)
Description: Weighted Sum of Pain Intensity Difference and Pain Relief Scores Over Six Hours (SPRID6) - pain intensity and pain relief were evaluated using a 0-100 mm visual analog scale (VAS) where 0 = no pain and 100 = very severe pain for pain intensity and 0 = no relief and 100 = complete relief for pain relief. For SPRID6, the total possible minimum value is -300 (worst) and the total possible maximum value is 1200 (best). The weights used in the calculation of weighted sums were equal to the elapsed time (hour) between the time point of interest and the preceding time point.
Time Frame: 6 Hours
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all subjects who were randomized, took study medication, did not vomit within 60 minutes after dosing, and had a baseline pain score and at least one post-randomization assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 529.4 (22.31) | 427.3 (22.21) | 60.0 (44.51)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; First test H1: acetaminophen 1000 mg vs placebo at the alpha = 0.025 one-tail level; If H1 was rejected then, Test H2: acetaminophen 1000 mg vs acetaminophen 650 mg, and Test H3: acetaminophen 650 mg vs placebo; H2 and H3 were each tested at the alpha = 0.025 one-tail level; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 469.37 — SPRID6 = 0.25 times (PRID at 15 min + PRID at 30 min + PRID at 45 min + PRID at 60 min + PRID at 75 min + PRID at 90 min) + 0.5 times (PRID at 120 minutes) + PRID at 3 hours + PRID at 4 hours + PRID at 5 hours + PRID at 6 hours
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, ANOVA; Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 102.09 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 367.28 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Sum of Pain Intensity Difference Over Six Hours (SPID6)
Description: Weighted Sum of the Pain Intensity Difference from Baseline Over Six Hours (SPID6) - pain intensity was evaluated using a 0-100 mm visual analog scale (VAS) where 0 = no pain and 100 = very severe pain. The total possible minimum value is -300 (worst) and the total possible maximum value is 600 (best). The weights used in the calculation of weighted sums were equal to the elapsed time (hour) between the time point of interest and the preceding time point.
Time Frame: 6 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 222.5 (10.49) | 174.3 (10.44) | -4.2 (20.93)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 226.70
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 48.14
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 178.56

3. Secondary Outcome: Sum of Pain Relief Scores Over Six Hours (TOTPAR6)
Description: Weighted Sum of the Pain Relief Scores Over Six Hours (TOTPAR6) - pain relief was evaluated using a 0-100 mm visual analog scale (VAS) where 0 = no relief and 100 = complete relief. The total possible minimum value is 0 (worst) and the total possible maximum value is 600 (best). The weights used in the calculation of weighted sums were equal to the elapsed time (hour) between the time point of interest and the preceding time point.
Time Frame: 6 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 306.9 (12.02) | 253.0 (11.96) | 64.3 (23.98)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 242.67
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.002, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 53.95
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 188.72

4. Secondary Outcome: Pain Intensity Difference (PID) at 15 Minutes
Description: Pain Intensity Difference (PID) from Baseline at Each Assessment Time point - pain intensity was evaluated using a 0-100 mm visual analog scale (VAS) where 0 = no pain and 100 = very severe pain with a highest possible score of 100. The pain intensity difference was calculated at each time point as the pain intensity score at baseline minus the pain intensity score at the stated time point.
Time Frame: 15 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 5.6 (0.92) | 6.9 (0.91) | 1.3 (1.83)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.037, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 4.30
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.294, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = -1.36
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.006, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 5.66

5. Secondary Outcome: Pain Intensity Difference (PID) at 30 Minutes
Description: as for outcome 4
Time Frame: 30 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 21.3 (1.48) | 21.5 (1.47) | 0.5 (2.95)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 20.85
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.946, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = -0.14
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 20.99

6. Secondary Outcome: Pain Intensity Difference (PID) at 45 Minutes
Description: as for outcome 4
Time Frame: 45 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 33.9 (1.71) | 32.8 (1.71) | 0.2 (3.42)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 33.68
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.661, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 1.06
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 32.62

7. Secondary Outcome: Pain Intensity Difference (PID) at 60 Minutes
Description: as for outcome 4
Time Frame: 60 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 40.4 (1.82) | 36.6 (1.81) | -0.1 (3.62)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 40.56
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.13, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 3.88
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 36.67

8. Secondary Outcome: Pain Intensity Difference (PID) at 75 Minutes
Description: as for outcome 4
Time Frame: 75 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 43.1 (1.88) | 37.6 (1.87) | -0.9 (3.74)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 43.97
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.041, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 5.42
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 38.55

9. Secondary Outcome: Pain Intensity Difference (PID) at 90 Minutes
Description: as for outcome 4
Time Frame: 90 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 44.4 (1.93) [1.92 to 3.85] | 38.0 (1.92) | -0.6 (3.85)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 44.97
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.02, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 6.34
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 38.63

10. Secondary Outcome: Pain Intensity Difference (PID) at 120 Minutes
Description: as for outcome 4
Time Frame: 120 Minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all subjects who were randomized, took study medication, and did not vomit within 60 minutes after dosing, had a baseline pain score and at least one post-randomization assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 44.8 (2.00) | 35.7 (1.99) | -2.7 (3.99)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 47.46
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 9.08
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 38.38

11. Secondary Outcome: Pain Intensity Difference (PID) at 180 Minutes
Description: as for outcome 4
Time Frame: 180 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 40.8 (2.03) | 31.9 (2.02) | -2.6 (4.05)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 43.42
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.002, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 8.83
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 34.59

12. Secondary Outcome: Pain Intensity Difference (PID) at 240 Minutes
Description: as for outcome 4
Time Frame: 240 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 40.8 (2.11) | 30.3 (2.10) | -1.1 (4.20)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 41.99
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 10.57
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 31.42

13. Secondary Outcome: Pain Intensity Difference (PID) at 300 Minutes
Description: as for outcome 4
Time Frame: 300 Minutes
Population: Analysis is based on the Intent-to-Treat (ITT) set, which included all subjects who were randomized, took study medication, and did not vomit within 60 minutes after dosing, and had a baseline pain score and at least one post-randomization assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 37.9 (2.17) | 27.1 (2.16) | -0.1 (4.32)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 38.04
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 10.82
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 27.22

14. Secondary Outcome: Pain Intensity Difference (PID) at 360 Minutes
Description: as for outcome 4
Time Frame: 360 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 33.4 (2.19) | 23.8 (2.18) | 1.0 (4.37)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 32.45
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.002, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 9.58
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 22.87

15. Secondary Outcome: Pain Relief (PAR) Scores at 15 Minutes
Description: Pain Relief Scores at each Assessment Timepoint - pain relief was evaluated using a 0-100 mm visual analog scale (VAS) where 0 = no relief and 100 = complete relief with a highest possible score of 100
Time Frame: 15 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 8.3 (1.09) | 9.4 (1.09) | 3.0 (2.18)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.028, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 5.35
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.462, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = -1.13
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.008, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 6.48

16. Secondary Outcome: Pain Relief (PAR) Scores at 30 Minutes
Description: as for outcome 15
Time Frame: 30 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 29.6 (1.84) | 29.9 (1.83) | 4.8 (3.66)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 24.81
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.907, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = -0.30
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 25.11

17. Secondary Outcome: Pain Relief (PAR) Scores at 45 Minutes
Description: as for outcome 15
Time Frame: 45 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 46.1 (2.10) | 44.8 (2.09) | 7.9 (4.18)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 38.19
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.655, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 1.32
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 36.87

18. Secondary Outcome: Pain Relief (PAR) Scores at 60 Minutes
Description: as for outcome 15
Time Frame: 60 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 54.4 (2.16) | 50.1 (2.15) | 8.3 (4.30)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 46.15
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.155, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 4.33
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 41.82

19. Secondary Outcome: Pain Relief (PAR) Scores at 75 Minutes
Description: as for outcome 15
Time Frame: 75 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 58.0 (2.18) | 52.0 (2.17) | 8.4 (4.35)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 49.69
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 6.04
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 43.65

20. Secondary Outcome: Pain Relief (PAR) Scores at 90 Minutes
Description: as for outcome 15
Time Frame: 90 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 59.9 (2.22) | 53.1 (2.21) | 10.1 (4.43)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 49.83
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.032, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 6.74
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 43.10

21. Secondary Outcome: Pain Relief (PAR) Scores at 120 Minutes
Description: as for outcome 15
Time Frame: 120 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 60.3 (2.25) | 50.8 (2.24) | 8.0 (4.49)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 52.36
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.003, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 9.52
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 42.84

22. Secondary Outcome: Pain Relief (PAR) Scores at 180 Minutes
Description: as for outcome 15
Time Frame: 180 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 56.3 (2.31) | 46.3 (2.30) | 9.5 (4.61)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 46.80
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.002, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 10.04
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 36.75

23. Secondary Outcome: Pain Relief (PAR) Scores at 240 Minutes
Description: as for outcome 15
Time Frame: 240 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 56.2 (2.41) | 44.3 (2.40) | 12.3 (4.81)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 43.84
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 11.82
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 32.02

24. Secondary Outcome: Pain Relief (PAR) Scores at 300 Minutes
Description: as for outcome 15
Time Frame: 300 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 52.2 (2.49) | 40.5 (2.48) | 13.8 (4.97)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 38.40
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 11.68
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 26.72

25. Secondary Outcome: Pain Relief (PAR) Scores at 360 Minutes
Description: as for outcome 15
Time Frame: 360 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 48.0 (2.51) | 36.6 (2.50) | 14.0 (5.02)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 33.94
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 11.40
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 22.55

26. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 15 Minutes
Description: Sum of PID and PAR Scores (PRID) at each Assessment Time point - pain intensity and pain relief were evaluated using a 0-100 mm visual analog scale (VAS) where 0 = no pain and 100 = very severe pain for pain intensity and 0 = no relief and 100 = complete relief for pain relief
Time Frame: 15 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 13.9 (1.95) | 16.4 (1.94) | 4.2 (3.89)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.027, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 9.65
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.365, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = -2.49
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.005, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 12.14

27. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 30 Minutes
Description: as for outcome 26
Time Frame: 30 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 50.9 (3.26) | 51.3 (3.24) | 5.2 (6.50)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 45.65
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.923, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = -0.45
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 46.10

28. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 45 Minutes
Description: as for outcome 26
Time Frame: 45 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 80.0 (3.76) | 77.6 (3.74) | 8.1 (7.49)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 71.87
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.653, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 2.38
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 69.49

29. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 60 Minutes
Description: as for outcome 26
Time Frame: 60 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 94.9 (3.92) | 86.7 (3.90) | 8.2 (7.81)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 86.71
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.138, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 8.21
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 78.49

30. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 75 Minutes
Description: as for outcome 26
Time Frame: 75 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 101.1 (4.00) | 89.6 (3.99) | 7.4 (7.99)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 93.66
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.043, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 11.46
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 82.20

31. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 90 Minutes
Description: as for outcome 26
Time Frame: 90 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 104.2 (4.10) | 91.2 (4.08) | 9.4 (8.18)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 94.80
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.024, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 13.08
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 81.72

32. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 120 Minutes
Description: as for outcome 26
Time Frame: 120 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 105.1 (4.20) | 86.5 (4.18) | 5.3 (8.38)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 99.82
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.002, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 18.60
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 81.23

33. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 180 Minutes
Description: as for outcome 26
Time Frame: 180 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 97.1 (4.29) | 78.2 (4.27) | 6.9 (8.56)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 90.22
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.002, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 18.87
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 71.35

34. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 240 Minutes
Description: as for outcome 26
Time Frame: 240 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 97.0 (4.47) | 74.6 (4.46) | 11.2 (8.93)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 85.82
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 22.39
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 63.44

35. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 300 Minutes
Description: as for outcome 26
Time Frame: 300 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 90.1 (4.62) | 67.6 (4.60) | 13.7 (9.22)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 76.44
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 22.50
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 53.94

36. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief Scores (PRID) at 360 Minutes
Description: as for outcome 26
Time Frame: 360 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
units on a scale | 81.4 (4.66) | 60.4 (4.64) | 15.0 (9.31)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 66.39
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.002, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 20.98
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 45.41

37. Secondary Outcome: Time to Meaningful Pain Relief
Description: Minutes until meaningful pain relief was achieved. A stopwatch was provided to the subject after ingestion of the study medication. The subject was instructed to stop the stopwatch when the relief from the starting pain was meaningful to them.
Time Frame: within 6 Hours
Population: as for outcome 1
Measure: Median (Full Range); unit: Minutes
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 238 | 241 | 60
Minutes | 53.7 [9.3 to 360] | 56.1 [15.9 to 360] | NA [NA to NA] — Data for the placebo group are not available. Median was not estimable since fewer than 50% of the subjects treated with Placebo obtained meaningful pain relief.
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Wilcoxon test, from SAS PROC LIFETEST — The significance threshold level was 0.05 (two-sided). p-Values are based on the Wilcoxon test from PROC LIFETEST that compared survival curves
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.26, Wilcoxon test, from SAS PROC LIFETEST — [p-value comment as in outcome 37, analysis 1]
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Wilcoxon test, from SAS PROC LIFETEST — [p-value comment as in outcome 37, analysis 1]

38. Secondary Outcome: Time to Confirmed Perceptible Pain Relief
Description: Minutes until confirmed perceptible pain relief was achieved. A stopwatch was provided to the subject after ingestion of the study medication. The subject was instructed to stop the stopwatch when they first began to feel any pain relieving effect whatsoever of the drug, that was when they first felt any pain relief. It did not necessarily mean they felt completely better, although they might have, but when they first felt any difference in the pain.
Time Frame: within 6 Hours
Population: as for outcome 1
Measure: Median (Full Range); unit: Minutes
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
Minutes | 22.2 [3.8 to 360] | 22.2 [3.8 to 360] | NA [NA to NA] — Data for the placebo group are not available. Median was not estimable because fewer than 50% of the subjects treated with Placebo obtained perceptible pain relief.
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Wilcoxon test, from SAS PROC LIFETEST — [p-value comment as in outcome 37, analysis 1]
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.934, Wilcoxon test, from SAS PROC LIFETEST — [p-value comment as in outcome 37, analysis 1]
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Wilcoxon test, from SAS PROC LIFETEST — [p-value comment as in outcome 37, analysis 1]

39. Secondary Outcome: Duration of Analgesia - Time to Rescue
Description: Minutes until rescue medication was given.
Time Frame: within 6 Hours
Population: as for outcome 1
Measure: Median (Full Range); unit: Minutes
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
Minutes | NA [NA to NA] — Data for the acetaminophen 1000 mg group are not available. Median was not estimable since fewer than 50% of the subjects treated with acetaminophen 1000 mg rescued. | NA [NA to NA] — Data for the acetaminophen 650 mg group are not available. Median was not estimable since fewer than 50% of the subjects treated with acetaminophen 650 mg rescued. | 99.5 [92 to 360]
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups. Subjects not rescuing during the 6-hour study period had their time to rescue set to 6 hours and were censored; Test type: Superiority or Other; p < 0.001, Log Rank — The significance threshold level was 0.05 (two-sided). p-Values are based on the log-rank test from PROC LIFETEST that compared survival curves
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; [analysis description as in outcome 39, analysis 1]; Test type: Superiority or Other; p < 0.001, Log Rank — [p-value comment as in outcome 39, analysis 1]
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; [analysis description as in outcome 39, analysis 1]; Test type: Superiority or Other; p < 0.001, Log Rank — [p-value comment as in outcome 39, analysis 1]

40. Secondary Outcome: Rescue Rates Through Four Hours
Description: Percentage of subjects using rescue medication.
Time Frame: through 4 Hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
Percentage of Participants | 20.1 | 32.4 | 80.0
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Stratified by categorical baseline pain rating; Odds Ratio (OR) = 0.06
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Stratified by categorical baseline pain rating; Odds Ratio (OR) = 0.52
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Stratified by categorical baseline pain rating; Odds Ratio (OR) = 0.12

41. Secondary Outcome: Rescue Rates Through Six Hours
Description: Percentage of subjects using rescue medication.
Time Frame: through 6 Hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
Percentage of Participants | 29.3 | 45.6 | 80.0
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Stratified by categorical baseline pain rating; Odds Ratio (OR) = 0.10
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Stratified by categorical baseline pain rating; Odds Ratio (OR) = 0.49
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Stratified by categorical baseline pain rating; Odds Ratio (OR) = 0.21

42. Secondary Outcome: Percentage of Subjects With >50% of the Maximum Possible TOTPAR6 Score
Description: Percentage of Subjects with >50% of the Maximum Possible TOTPAR6 Score - pain relief was evaluated using a 0-100 mm visual analog scale (VAS) where 0 = no relief and 100 = complete relief with a highest possible score of 600 so >50% is >300 out of 600
Time Frame: 6 Hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
Percentage of Participants | 56.9 | 44.4 | 6.7
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Stratified by categorical baseline pain rating; Odds Ratio (OR) = 18.45
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Stratified by categorical baseline pain rating; Odds Ratio (OR) = 1.65
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The significance threshold level was 0.05 (two-sided); Stratified by categorical baseline pain rating; Odds Ratio (OR) = 11.16

43. Secondary Outcome: Patient Global Evaluation
Description: Patient Assessment of the Pain Medication - Number of Subjects rating the medication they received as a pain reliever on a score of 0-4, where 0=poor, 1=fair, 2=good, 3=very good, 4=excellent
Time Frame: 6 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Number analyzed (Participants) | 239 | 241 | 60
Units on a scale | 2.28 (0.073) | 1.95 (0.073) | 0.60 (0.146)
Statistical Analysis 1: Comparison: ACE-1000 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 1.68
Statistical Analysis 2: Comparison: ACE-1000 vs ACE-650; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 0.33
Statistical Analysis 3: Comparison: ACE-650 vs ACE-0; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p < 0.001, ANOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline pain categorical ratings were factors; Mean Difference (Final Values) = 1.35

ADVERSE EVENTS:
Time Frame: 6 Hours (+30 days for Serious Adverse Events)
Description: The safety analysis set included all subjects who were randomized and took study medication.
Arm/Group | ACE-1000 | ACE-650 | ACE-0
Serious Adverse Events (participants affected / at risk) | 0/239 | 0/241 | 0/60
Other Adverse Events (participants affected / at risk) | 45/239 | 42/241 | 13/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACE-1000 (N=239) | ACE-650 (N=241) | ACE-0 (N=60)
Nausea (Gastrointestinal disorders) | 29 | 26 | 9
Vomiting (Gastrointestinal disorders) | 11 | 11 | 4
Dizziness (Nervous system disorders) | 10 | 8 | 4

LIMITATIONS AND CAVEATS:
Analysis is based on the Intent-to-Treat (ITT) set, which included all subjects who were randomized, took study medication, did not vomit within 60 minutes after dosing, and had a baseline pain score and at least one post-randomization assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results may not be published or referred to at research seminars, lectures or professional meetings, in whole or in part, without the prior written consent of McNeil Consumer Healthcare, to be given or withheld at McNeil Consumer Healthcare's sole and absolute discretion